CLINICAL TRIAL: NCT07406997
Title: Rehabilitation With Empowered STrategies to Optimize REcovery After Spine Surgery
Brief Title: Rehabilitation With Empowered STrategies to Optimize REcovery
Acronym: RESTORE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kristin Archer, Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 251516; HT9425-25-1-0925 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Lumbar Spine Degenerative Changes; Lumbar Spine Surgery
Keywords: behavioral research; Patient Reported Outcomes Measures; Pain; Pain Catastrophizing
MeSH Terms: conditions — Pain | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empowered Relief (Experimental): Remotely delivered group session with behavioral strategies
  Interventions: Behavioral: Empowered Relief
- Education (Active Comparator): Remotely delivered group session with educational information
  Interventions: Other: Education

INTERVENTIONS:
Behavioral: Empowered Relief — Empowered Relief (ER) is a single-session group class that has two main components of pain neuroscience education and pain coping skills based on cognitive-behavioral principles.
  Arms: Empowered Relief
Other: Education — Education program is a single-session group class that includes information on how to manage pain and disability, prevent future injury and stay healthy after back surgery.
  Arms: Education

SUMMARY:
The main goal of this clinical trial is to understand the benefits of remotely delivered Empowered Relief in patients undergoing lumbar spine surgery. The main question the trial aims to answer is:

Does a postoperative behavioral intervention, Empowered Relief, performed early after back surgery have a measurable impact on postoperative outcomes?

Additional questions are whether changes in pain catastrophizing are related to improvements in outcomes and whether preoperative pain catastrophizing is a moderator of response to treatment.

Researchers will compare remotely delivered Empowered Relief to remotely delivered education to see if Empowered Relief helps patients manage their pain and functional limitations after back surgery.

Participants will:

* Complete one group session of remotely delivered Empowered Relief or Education after back surgery
* Complete surveys before surgery and 3- and 6-months after surgery

DETAILED DESCRIPTION:
The proposed study will conduct a phase II, two-group randomized controlled trial in patients undergoing lumbar spine surgery. Patients will be enrolled and randomized prior to spine surgery from a civilian medical center and military treatment facilities. Patients will be randomized to either (1) 1-session Empowered Relief or (2) 1-session Education. Both interventions are delivered remotely in a group setting through a web-based platform by licensed health care professionals. Outcome assessments will be conducted by evaluators blinded to group assignment at 3-months and 6-months after surgery.The results of our clinical trial will advance research on remote nonpharmacologic strategies for managing pain and improving quality of life post-surgery in both civilian and military patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Surgical treatment of a lumbar degenerative condition using a laminectomy with or without fusion procedure
* English speaking
* Age between 18-75 years

Exclusion Criteria:

* Surgery due to trauma, fracture, tumor, infection, or spinal deformity
* Revision surgery
* Prior history of lumbar spine surgery in last 5 years
* Involved in litigation or a workers' compensation claim due to injury
* Currently undergoing treatment for cancer
* Unable to access a reliable internet connection
* Unable to provide a stable telephone or physical address
* Unable to participate in follow-up assessment for 6 months after surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-11 (Estimated); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Pain Interference | 3 and 6 months after hospital discharge
  PROMIS Pain Interference domain

SECONDARY OUTCOMES:
Physical Function | 3 and 6 months after hospital discharge
  PROMIS Physical Function Domain
Disability | 3 and 6 months after hospital discharge
  Oswestry Disability Index
Pain Intensity | 3 and 6 months after hospital discharge
  Numeric Rating Scale for back pain and leg pain
Opioid Use | 3 and 6 months after hospital discharge
  morphine milligram equivalents

OTHER OUTCOMES:
Pain Catastrophizing | 3 and 6 months after hospital discharge
  Pain Catastrophizing Scale
Sleep | 3 and 6 months after hospital discharge
  PROMIS Sleep Disturbance domain
Patient Satisfaction | 3 and 6 months after hospital discharge
  NASS Patient Satisfaction Index
Employment | 3 and 6 months after hospital discharge
  Return to work or duty and date of return

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Madigan Army Medical Center, Joint Base Lewis McChord, Washington

IPD SHARING:
Plan to Share IPD: No